CLINICAL TRIAL: NCT01929343
Title: Lidocaine Infusion as a Treatment for Cocaine Relapse and Craving
Acronym: LIDO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bryon Adinoff (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Bryon Adinoff, Clinical Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU 032013-049
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Cocaine Addiction
Keywords: cocaine; addiction; lidocaine; memory; drug abuse
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive; Substance-Related Disorders | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- lidocaine following cue-induced craving (Experimental): Lidocaine will be administered immediately following craving induction. Lidocaine will administered at a loading dose of 2mg/kg(milligrams per kilogram) initial bolus over 5 minutes lidocaine followed by continuous infusion at 2mg/kg /hour for 4 hours.
  Interventions: Drug: lidocaine following cue-induced craving
- lidocaine following neutral stimulus (Active Comparator): Lidocaine will be administered immediately following neutral stimulus. Lidocaine will administered at a loading dose of 2mg/kg initial bolus over 5 minutes lidocaine followed by continuous infusion at 2mg/kg /hour for 4 hours.
  Interventions: Drug: lidocaine following neutral stimulus
- saline (Placebo Comparator): Saline will be administered at same volume of lidocaine in active arms.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: lidocaine following cue-induced craving — as described in Arm Description
  Other Names: Xylocaine
  Arms: lidocaine following cue-induced craving
Drug: lidocaine following neutral stimulus — as described in Arm Description
  Other Names: Xylocaine
  Arms: lidocaine following neutral stimulus
Drug: saline — as described in Arm Description
  Other Names: 0.9% Sodium chloride
  Arms: saline

SUMMARY:
We propose that the systemic administration of lidocaine following the induction of cue-induced craving, relative to saline plus cue-induced craving or lidocaine without cue-induced craving, will block the reconsolidation of cue memories. This will lead to a reduction in cue-induced craving upon repeated testing as well as subsequent cocaine use and basal craving.

DETAILED DESCRIPTION:
Cocaine dependence is among the most tenacious of the substance use disorders yet remains one of the few lacking an effective pharmacological intervention. As other pharmacologic approaches have not been fruitful, new targets are required. A novel treatment approach is to disrupt the neural processes involved in cue-related memories (memory links between the external stimuli associated with drug use and the subjective drug effect). These engrained memories, when reactivated by cues, elicit craving and a return to drug use. Each cue re-exposure, however, requires the re-remembering (or reconsolidation) of the drug cue. Key molecular processes required for memory reconsolidation are NMDA (N-methyl-D-aspartate) receptor activation, the induction of nitric oxide (NO) synthesis and increased extracellular signal-regulated kinase (ERK) activity. In rodent models, blocking these processes changes the cue-related memory; the cue loses its potency to induce a return to drug self-administration. Lidocaine is an FDA (Food and Drug Administration) approved medication that inhibits activation of NMDA (N-methyl-D-aspartate) receptors and suppresses production of NO (nitric oxide) and ERK (extracellular signal-regulated kinase). Lidocaine, like cocaine, is a local anesthetic with potent effects as a sodium-channel blocker. Unlike cocaine, lidocaine is essentially devoid of activity at monoamine re-uptake transporters and has no rewarding or addictive properties. As lidocaine suppresses the molecular processes required for drug cue reconsolidation and has relatively specific effects upon the striatal regions necessary for drug cue reconsolidation, lidocaine may offer a novel approach for interfering with memory reconsolidation. Two other (Sodium) Na+ channel blockers have also decrease craving and/or substance use in substance-dependent subjects. We propose that the systemic administration of lidocaine following the induction of cue-induced craving, relative to saline plus cue-induced craving or lidocaine without cue-induced craving, will block the reconsolidation of cue memories. This will lead to a reduction in cue-induced craving upon repeated testing as well as subsequent cocaine use and basal craving. If our hypotheses are proven correct, these findings will 1) support a role for lidocaine in cocaine addiction treatment, 2) demonstrate the feasibility and efficacy of attenuating cue-induced memories, and 3) guide the development of a larger study with lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* 25-60 years old
* men or women
* any race or ethnicity
* cocaine addition is primary present and lifetime drug of abuse
* live locally

Exclusion Criteria:

* Patients with active DSM (Diagnostic Statistical Manual)-IV other Substance Dependence (except nicotine) within the previous three months, Affective Disorder, Schizophrenic Disorders.
* significant cognitive impairment (WTAR<70) (Wechsler Test of Adult Reading <70)..
* use of tricyclic anti-depressants, benzodiazepines, cimetidine, mood stabilizers, opioids, lithium, sympathomimetics, anticonvulsants, sedative/hypnotics, β-blockers, or dopamine agonists will be excluded from the study.
* Medical conditions that might limit cooperation (e.g. dementia) or put the patient at medical risk (i.e. significant hematologic, hepatic, renal, or cardiovascular pathology - particularly arrhythmias) will be excluded.
* Patients with congenital or idiopathic methemoglobinemia or patients taking medications associated with increased risk of methemoglobinemia (including sulfonamides, acetaminophen, acetanilid, aniline dyes, benzocaine, chloroquine, dapsone, naphthalene, nitrates and nitrites, nitrofurantoin, nitroglycerin, nitroprusside, pamaquine, paraaminosalicylic acid, phenacetin, phenobarbital, phenytoin, primaquine, quinine) will be excluded.
* Patients with past or present neurologic disorders (i.e. severe head trauma, transient ischemic attacks, stroke, tumor, etc.) will be excluded. - Active suicidal ideation, pregnant or nursing women, and prisoners will be excluded from the study.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryon Adinoff, MD, Principal Investigator — UT Southwestern Medical Center, VA North Texas Health Care System
Locations (1):
- UT Southwestern Medical Center at Dallas, Division on Addictions, Dallas, Texas, United States

REFERENCES:
- [Derived] Becker JE, Price JL, Leonard D, Suris A, Kandil E, Shaw M, Kroener S, Brown ES, Adinoff B. The Efficacy of Lidocaine in Disrupting Cocaine Cue-Induced Memory Reconsolidation. Drug Alcohol Depend. 2020 Jul 1;212:108062. doi: 10.1016/j.drugalcdep.2020.108062. Epub 2020 May 12. PMID 32480252

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 84 participants were consented to participate in the study. 48 were withdrawn as they did not meet inclusion/exclusion criteria (insufficient use of cocaine, medical concerns, positive drug screens or psychiatric disorders) upon further screening and evaluation. Thus, we are reporting on 36 participants.
Groups:
- Lidocaine Following Cue-induced Craving: Lidocaine will be administered immediately following craving induction. Lidocaine will administered at a loading dose of 2mg/kg initial bolus over 5 minutes lidocaine followed by continuous infusion at 2mg/kg /hour for 4 hours.
  lidocaine following cue-induced craving: as described in Arm Description
Period: Overall Study
Arm/Group | Lidocaine Following Cue-induced Craving | Lidocaine Following Neutral Stimulus | Saline
Started | 12 | 9 | 12
Completed | 11 | 7 | 12
Not Completed | 1 | 2 | 0
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine Following Cue-induced Craving | Lidocaine Following Neutral Stimulus | Saline | Total
Number analyzed (Participants) | 12 | 9 | 12 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 9 | 12 | 33
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 8
  Male | 9 | 7 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Cue-induced Craving After Lidocaine/Saline Administration.
Description: 7 days after lidocaine/saline administration, cocaine craving will be measured during the administration of relaxation or craving script. Craving intensity will be measured by the subjective intensity of craving as reported by the participant. Measured via a visual analog scale based on 4 (out of 10) questions from the Cocaine Craving Questionnaire (1-strongly disagree to 7- strongly agree). Highest total score possible 28, lowest score possible is 4. If the score is low in the lidocaine group and high in the saline group, it would mean that lidocaine has successfully decreased the craving response relative to saline.
Time Frame: craving measured immediately following reading of the script.
Population: 3 participants were lost to follow-up and hence we could analyze only the available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine Following Cue-induced Craving | Lidocaine Following Neutral Stimulus | Saline
Number analyzed (Participants) | 11 | 7 | 12
units on a scale | 31.7 (12.6) | 17.3 (9.5) | 22.7 (11.9)

2. Primary Outcome: Physiological Responses as Measured by Heart Rate After Lidocaine/Saline Administration.
Description: 7 days after lidocaine/saline administration, heart rate will be measured during the administration of a relaxation or craving script. Heart rate will be measured in beats per minute.
Time Frame: 120 seconds, during reading of the script.
Population: 3 participants were lost to follow-up and hence we could analyze only the available data.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Lidocaine Following Cue-induced Craving | Lidocaine Following Neutral Stimulus | Saline
Number analyzed (Participants) | 11 | 7 | 12
beats per minute | 67.4 (27.4) | 73.0 (19.4) | 77.5 (16.6)

3. Primary Outcome: Physiological Responses as Measured by Blood Pressure After Lidocaine/Saline Administration.
Description: 7 days after lidocaine/saline administration, blood pressure (BP) response will be assessed during relaxation or craving script. Blood pressure will be measured by mmHg.
Time Frame: BP will measured during the two minutes of script reading.
Population: The data was not collected and hence was not analyzed.
Arm/Group | Lidocaine Following Cue-induced Craving | Lidocaine Following Neutral Stimulus | Saline
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Physiological Responses as Measured by Galvanic Skin Response (GSR) After Lidocaine/Saline Administration.
Description: 7 days after lidocaine/saline administration, GSR will be measured during the reading of the relaxation or saline script. It is predicted that higher GSR would be associated with higher cocaine craving and lower GSR will be associated with lower cocaine craving.
Time Frame: 2 minutes during script reading.
Population: 3 participants were lost to follow-up and hence we could analyze only the available data.
Measure: Mean (Standard Deviation); unit: EDA Amplitute (uS)
Arm/Group | Lidocaine Following Cue-induced Craving | Lidocaine Following Neutral Stimulus | Saline
Number analyzed (Participants) | 11 | 7 | 12
EDA Amplitute (uS) | 19.1 (4.5) | 20.1 (0.2) | 20.4 (0.7)

5. Primary Outcome: Physiological Responses as Measured by EMG (Electromyography) After Lidocaine/Saline Administration.
Description: Electromyography (frontal) will be measured during the administration of the relaxation or craving script seven days after infusion. EMG is assessed by uV (microvolts). Higher scores reflect greater amounts of EMG activity, lower scores reflect lower amounts of EMG activity. It was expected that EMG would be positively associated with cocaine craving.
Time Frame: 2 minutes during administration of script.
Measure: Mean (Standard Deviation); unit: uV
Arm/Group | Lidocaine Following Cue-induced Craving | Lidocaine Following Neutral Stimulus | Saline
Number analyzed (Participants) | 10 | 7 | 12
uV | 21.6 (44.5) | 28.1 (57.8) | 5.9 (2.1)

6. Secondary Outcome: Cocaine Use
Description: cocaine use will be measured by urine drug screen and participant self-report three times weekly after lidocaine/saline administration. Cocaine use will be assessed as positive (1) or negative (0) using urine drug screen for cocaine and/or by participant self-report of cocaine use.
Time Frame: cocaine use will be measure during the 4 weeks following infusion
Measure: Mean (Standard Deviation); unit: days of cocaine used/week
Arm/Group | Lidocaine Following Cue-induced Craving | Lidocaine Following Neutral Stimulus | Saline
Number analyzed (Participants) | 10 | 7 | 11
days of cocaine used/week | 3.8 (1.8) | 2.7 (0.8) | 3.0 (0.0)

7. Secondary Outcome: Cocaine Craving
Description: basal measures of cocaine craving will be measured by Cocaine Craving Questionnaire (CCQ) times weekly after lidocaine/saline administration. The higher the score the more craving and lower the score the less craving. The CCQ has 10 items, each item scored 1-7. Maximum score is 70, minimum score is 7.
Time Frame: cocaine craving will be measure during the 4 weeks following infusion
Population: Only available data were analyzed. Some participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine Following Cue-induced Craving | Lidocaine Following Neutral Stimulus | Saline
Number analyzed (Participants) | 11 | 7 | 12
units on a scale | 32.3 (18.5) | 15.8 (4.8) | 20.9 (15.6)

ADVERSE EVENTS:
Time Frame: 4 weeks following lidocaine/saline administration
Arm/Group | Lidocaine Following Cue-induced Craving | Lidocaine Following Neutral Stimulus | Saline
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/12

LIMITATIONS AND CAVEATS:
Within the Primary outcome measure- 'Physiological Responses as Measured by Blood Pressure After Lidocaine/Saline Administration', we're unable to report this as it was not actually an outcome of interest and so was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT01929343/Prot_SAP_000.pdf